CLINICAL TRIAL: NCT02681718
Title: Controlling Hyperglycemia Among Minority Population (CHAMP): A Randomized Controlled Trial of Two Diabetes Interventions for Underserved Communities
Brief Title: Controlling Hyperglycemia Among Minority Population
Acronym: CHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai Health System (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSH15-46
Record Dates: First submitted 2016-02-03; First posted 2016-02-12 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Diabetes
Keywords: A1C≥9%; minorities; economically disadvantaged
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Community Health Worker education (Experimental): During a six-month intervention period, the CHWs will conduct six home-based visitations and provide individualized diabetes education using an intensive diabetes lifestyle curriculum called Diabetes Learning Circle (DLC), developed and used by the Sinai Diabetes Education Program. At each visit, lasting for approximately one hour, the participants will be motivated to set SMART behavioral goals for diabetes self-management. At each visit after the initial visit, CHWs will follow-up with each participant to check their progress on their behavioral SMART goals. In addition, the CHWs will conduct intermittent phone calls (at least one monthly) and home visits as needed.
  Interventions: Behavioral: Community health worker education
- Cell phone text messaging (Experimental): The participants in the text messaging group will receive weekly text messages through CareMessage. Each participant will receive 3-4 text messages per week for 6 months.
  Interventions: Behavioral: Cell phone text messaging
- Control (No Intervention): The participants in the control group will receive education as determined by the hospital's diabetes educator, dietitian, physician, or the participant's managed care provider. No additional education will be provided by the research team.

INTERVENTIONS:
Behavioral: Community health worker education — Diabetes self-management education by community health workers
  Arms: Community Health Worker education
Behavioral: Cell phone text messaging — Diabetes self-management education through cell phone text messaging
  Arms: Cell phone text messaging

SUMMARY:
The purpose of this study is to compare the efficacy of three approaches in diabetes management: (1) community health worker (CHW) education; (2) text messaging; and (3) usual hospital-based care. The goal is to determine the most cost-effective method of diabetes management among an economically-disadvantaged, minority population.

DETAILED DESCRIPTION:
The CHAMP study will test the efficacy of two interventions designed to decrease uncontrolled hyperglycemia (defined as Hemoglobin-A1C (A1C) at or above 9%) among adults with diabetes. Patients from a safety-net hospital will be randomized into three groups: 1) a control group, 2) an intervention providing diabetes self-care text messages, or 3) an intervention using community health workers to provide diabetes education and linkage to care. Secondary objectives include increasing diabetes knowledge, improving diabetes self-management, and increasing use of primary care (i.e., make one visit to the physician in 6 months) among the intervention participants. A cost-effectiveness analysis will determine the most appropriate way to reduce the burden of uncontrolled diabetes.

ELIGIBILITY:
Inclusion Criteria:

*Hyperglycemia with A1C ≥9%

Exclusion Criteria:

* Lives greater than 20 miles driving distance from Mount Sinai Hospital
* Pregnant women with gestational diabetes
* Advanced end-organ complications due to diabetes that include: end-stage renal disease, stroke with paresis, Congestive Heart Failure (NYHA class III or IV), or other major end-organ complication of diabetes
* Receiving treatment for a major psychiatric disorder (i.e. schizophrenia)
* Unable to understand and give informed consent in either English or Spanish
* Currently or previously participated in a diabetes research study
* Family member currently enrolled in a diabetes research study
* Previously received diabetes care related cell phone text messages
* Unable to receive text messages 3-4 times per week
* Living in a homeless shelter or temporary housing
* Plans to travel outside of the United States for more than 3 months in next year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Difference in Hemoglobin A1C (CHW vs. Control) | 6 months
  To assess whether there is a statistically significant difference in HbA1C level between CHW and control groups at 6 months follow-up.
Difference in Hemoglobin A1C (Text Message vs. Control) | 6 months
  To assess whether there is a statistically significant difference in HbA1C level between text message and control groups at 6 months follow-up.

SECONDARY OUTCOMES:
Percentage change in diabetes knowledge test scores | 6 months
  Michigan Diabetes and Research Center Knowledge test
Mean change in diabetes self-efficacy scores | 6 months
  Perceived competence in diabetes scale
Mean change in diabetes distress scores | 6 months
  Problem areas in diabetes (PAID-5) scale
Mean change in participants' beliefs about using insulin scores | 6 months
  Insulin treatment appraisal (ITAS) scale
Mean changes in diabetes self-care activities | 6 months
  Diabetes self-care activities include: diet, physical activity, self-monitoring of blood glucose, foot-care, and smoking
Percentage of participants who visited a physician due to a diabetes related follow-up | 6 months
  Self- reported

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No